CLINICAL TRIAL: NCT03649880
Title: Feasibility of [¹⁸F]-Fluoromisonidazole (FMISO) in Assessment of Malignant Brain Tumors
Brief Title: Feasibility of FMISO in Brain Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other); Weill Cornell University (Unknown)
Responsible Party: Principal Investigator, Ramon Barajas, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00016043; NCI-2018-01479 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00016043 (Other: OHSU Knight Cancer Institute); K08CA237809 (NIH)
Record Dates: First submitted 2018-08-06; First posted 2018-08-28 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Malignant Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — fluoromisonidazole; Magnetic Resonance Spectroscopy; Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (FMISO, PET/MRI or PET/CT) (Experimental): Participants receive FMISO intravenously (IV). Participants also undergo dynamic PET/computed tomography (CT) or PET/MRI over 120 minutes beginning 1 minute prior to FMISO injection, and static PET/CT or PET/MRI over 20-40 minutes approximately 90 minutes after FMISO injection. Participants then undergo a retest examination within 7 days. Participants may undergo 2 more PET/MRI or PET/CT scans no sooner than every 4 weeks. Supplemental oxygen may be administered to effect MRI signal.
  Interventions: Drug: ¹⁸F-Fluoromisonidazole; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Oxygen Therapy

INTERVENTIONS:
Drug: ¹⁸F-Fluoromisonidazole — Given IV
  Other Names: ¹⁸F-MISO; ¹⁸F-Misonidazole; FMISO
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI or PET/CT
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Procedure: Oxygen Therapy — Receive supplemental oxygen
  Other Names: supplemental oxygen therapy

SUMMARY:
This phase II trial studies how well ¹⁸F- fluoromisonidazole (FMISO) works with positron emission tomography (PET)/magnetic resonance imaging (MRI) in assessing participants with malignant (cancerous) brain tumors. FMISO provides information about the oxygen levels in a tumor, which may affect how the tumor behaves. PET/MRI imaging produces images of the brain and how the body functions. FMISO PET/MRI may help investigators see how much oxygen is getting in the brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of obtaining ¹⁸F- fluoromisonidazole (FMISO) PET (hypoxic volume and tumor to blood background values [T/B]) and dynamic susceptibility contrast enhanced (DSC) & diffusion-weighted imaging (DWI) MRI measures in patients with intracranial brain tumors.

II. Determine if MRI contrast-enhancement and hypoxic volume are imaging profiles of glioblastoma immunotherapy-mediated pseudoprogression or true progression in a clinical trial.

SECONDARY OBJECTIVE:

I. Determine the feasibility of baseline and follow-up FMISO PET and MR imaging co-registration.

TERTIARY OBJECTIVE:

I. Determine the reproducibility of the baseline FMISO PET imaging metrics as assessed by baseline "test" and "retest" experiments.

OUTLINE:

Participants receive FMISO intravenously (IV). Participants also undergo dynamic PET/computed tomography (CT) or PET/MRI over 120 minutes beginning 1 minute prior to FMISO injection, and static PET/CT or PET/MRI over 20-40 minutes approximately 90 minutes after FMISO injection. Participants then undergo a retest examination within 7 days. Participants may undergo 2 more PET/MRI or PET/CT scans no sooner than every 4 weeks. Supplemental oxygen may be administered to effect MRI signal.

After conclusion of the diagnostic tests, participants are followed for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (greater than 18 years of age) with a known or suspected intracranial tumor.
* Able to provide informed written consent and/or acceptable surrogate capable of providing consent on the patient's behalf.
* Legally authorized representative (LAR)-signed informed consent and assent obtained for those subjects identified as decisionally impaired
* Intracranial lesion known or suspected to be neoplastic greater than 10 mL as assessed by T2/fluid attenuated inversion recovery (FLAIR) MR imaging.
* Karnofsky performance score > 60 or Eastern Cooperative Oncology Group (ECOG) < 3 as assessed by referring clinician.
* Planning to undergo or previously received therapeutic intervention for the intracranial tumor.

Exclusion Criteria:

* Pregnant or breast feeding.
* Contraindication to PET, MRI, FMISO, or intravenous gadolinium based contrast agents.

  * Claustrophobia.
  * Weight greater than modality maximum capacity.
  * Presence of metallic foreign body or implanted medical devices in body not documented as MRI safe according to the Oregon Health & Science University (OHSU) Department of Radiology guidelines (including but not limited to cardiac pacemaker, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants).
  * Sickle cell disease.
  * Reduced renal function, as determined by glomerular filtration rate (GFR) < 45 mL/min/1.73 m^2 based on a serum creatinine level obtained per OHSU Department of Radiology and Advanced Imaging Research Center (AIRC) clinical criteria.
  * History of allergic reactions attributed to compounds of similar chemical or biologic composition to FMISO. An allergic reaction to nitroimidazoles is highly unlikely.
  * Unsure of pregnancy status as assessed by Department of Radiology and AIRC guidelines.
  * Subjects for whom supplemental oxygen could be harmful such as people with potential for hypoventilation (end-stage COPD, OSA on CPAP/Bi-PAP, etc).
  * Subjects with a relative contraindication to supplemental oxygen administration will not be provided oxygen but may still participate in the study.
* Presence of any other co-existing condition that, in the judgment of the principal investigator, might increase the risk to the subject (i.e., plans for hospice or end of life care).
* Poor peripheral intravenous access evaluated by patient history.
* Presence of other serious systemic illnesses, including: uncontrolled infection, other uncontrolled malignancy, uncontrolled diabetes type II, or psychiatric/social situations which might impact the endpoint of the study or limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Macro-imaging level feasibility | One day of diagnostic imaging
  Assessed as a factor of generating quantitative positron emission tomography (PET)/magnetic resonance imaging (MRI) metrics (intra-tumoral FMISO tumor to blood [T/B] level, hypoxic volume, dynamic susceptibility contrast enhanced [DSC], and diffusion-weighted imaging [DWI] values, and tissue oxygen maps). Images generated during the administration of oxygen will be used to generate tissue oxygen maps of the brain. Following completion of cohort enrollment, the generation of each quantitative PET/MRI metric will be independently scored as a dichotomous variable; successful or non-successful. Proportional assessment will be performed to assess for project feasibility. The successful generation of PET/MRI metrics in 85% of the initial cohort successfully imaged will need to be achieved for the imaging modality to be deemed feasible for this study. The estimated proportion of success rate for each metric along with the corresponding 95% binomial confidence interval will be provided.
MRI contrast enhancement | Up to 5 years
  Measured by Response assessment in neuro-oncology criteria sum product diameter assessment. The primary outcomes for this aim are enhancement mismatch ratio and hypoxic volume. Differences in imaging metrics will be evaluated using two sample t-test. If normal assumption is not satisfied, data transformation, or 95% confidence intervals based on bootstrapping method will be used. Exploratory analysis will assess diagnostic performance of imaging metrics (mismatch ratio and hypoxic volume) to identify pseudoprogression at earlier imaging dates.

SECONDARY OUTCOMES:
Technical feasibility of PET/MRI | Baseline to the start of long-term follow-up (up to 5 years)
  The generation of co-registered imaging data sets will be independently scored as a dichotomous variable; successful or non-successful (< 10mm versus [vs.] > 10mm alignment error). Proportional assessment will be performed to assess for project feasibility. The estimated proportion along with the corresponding 95% binomial confidence interval will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Barajas, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States